CLINICAL TRIAL: NCT06271395
Title: The Impact of Ultrasound-guided Botulinum Toxin Injection on Cricopharyngeal Muscle Dysfunction Under Balloon Localization
Brief Title: Ultrasound-guided Botulinum Toxin Injection on Cricopharyngeal Muscle Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Research Director, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chaoshengqiunang
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Cricopharyngeal Achalasia
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The observation group (Experimental): This group will be given Left cricopharyngeal muscle botulinum toxin injection, Injectable Type A Botulinum Toxin (National Medical Products Administration Approval Number S10970037) 100 unit, diluted with 1ml of 0.9% sodium chloride solution for injection and kept ready for use. Only once.
  Interventions: Drug: Injectable Type A Botulinum Toxin

INTERVENTIONS:
Drug: Injectable Type A Botulinum Toxin — Injectable Type A Botulinum Toxin (National Medical Products Administration Approval Number S10970037) 100 unit, diluted with 1ml of 0.9% sodium chloride solution for injection and kept ready for use. Only once. Using an ultrasound probe to scan the neck, the position of the lowest point, highest point, and lower middle point of the esophageal high-pressure zone are determined, and marks are made on the body surface and catheter wall. The high-pressure point and the lower middle point are selected as injection sites on the left side. The above area is locally disinfected, and the probe is covered with a sterile cover and coated with sterile coupling agent. Using a plane approach, 0.3ml or 30 unit of botulinum toxin is injected separately after reaching the esophageal circular layer at each of the two left injection points. A total of 60 unit of botulinum toxin is injected at the two left points.
  Other Names: Botulinum Toxin Injection

SUMMARY:
Ultrasound-guided injection is a visual, convenient, and radiation-free technique that allows real-time observation of the needle insertion process and drug injection location. The combination with a balloon for fixation further enhances the precision of the injection. In this study, we employed ultrasound-guided injection combined with balloon localization for cricopharyngeal muscle botulinum toxin injection treatment and conducted clinical observations.

DETAILED DESCRIPTION:
The patient's long-term inadequate food intake leads to malnutrition, decreased quality of life, and impacts the prognosis of the disease. Currently, both domestically and internationally, treatment options for cricopharyngeal muscle dysfunction include balloon dilation technique, surgical incision, and botulinum toxin injection. Passive dilation with a balloon can easily cause mucosal edema and damage. Cricopharyngeal myotomy surgery often presents complications such as local infection, excessive bleeding, and local nerve damage. Botulinum toxin can alleviate muscle spasms and has been widely used in the treatment of hypertonic disorders [3]. Common injection localization methods include ultrasound, electromyography, and endoscopy. Ultrasound-guided injection is a visual, convenient, and radiation-free technique that allows real-time observation of the needle insertion process and drug injection location. Combining it with balloon fixation further enhances the precision of the injection. In this study, we employed ultrasound-guided injection combined with balloon localization for cricopharyngeal muscle botulinum toxin injection treatment and conducted clinical observations.

ELIGIBILITY:
Inclusion Criteria:

* Videofluoroscopic swallowing study (VFSS) confirming incomplete/opening dysfunction of the cricopharyngeal muscle;
* No significant improvement in swallowing function after standardized rehabilitation treatment for more than 2 weeks (unchanged or decreased FOIS);
* Presence of swallowing initiation, with VFSS showing that the upward movement of the hyoid bone during swallowing is greater than half the height of the C3 vertebral body;
* Stable vital signs, alert consciousness, and cooperation with treatment;

Exclusion Criteria:

* Patients with severe cognitive impairments, psychiatric disorders, and severe cardiopulmonary diseases;
* Abnormalities in the pharynx and larynx structures;
* Patients with malignant tumors;
* Patients with infections or wounds at the injection site;
* Patients allergic to botulinum toxin; Patients with bleeding tendencies or coagulation disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
functional oral intake scale | day 1, day 15, day 29, day 169
  The Functional Oral Intake Scale (FOIS) is a tool used to assess the functional oral intake of individuals with dysphagia. The scale ranges from Level 1 to Level 7, with Level 1 indicating nothing by mouth and Level 7 representing total oral diet with no restrictions. In this scale, a higher score indicates better functional oral intake capabilities, meaning that higher levels correspond to better oral intake abilities.

SECONDARY OUTCOMES:
Penetration-Aspiration Scale | day 1, day 15, day 29, day 169
  The Penetration-Aspiration Scale (PAS) is a tool used to evaluate the severity of penetration and aspiration events that occur during swallowing. It assesses the extent to which food or liquid enters the airway during swallowing, indicating potential risks to respiratory health.
  The PAS ranges from Level 1 to Level 8, with Level 1 representing no penetration or aspiration and Level 8 representing material entering the airway with no effort to eject it. In this scale, a lower score indicates better swallowing function, as lower levels indicate less penetration or aspiration occurring during the swallowing process. It is important to minimize penetration and aspiration events to reduce the risk of respiratory complications and maintain optimal swallowing function.
The Fiberoptic Endoscopic Dysphagia Severity Scale | day 1, day 15, day 29, day 169
  The Fiberoptic Endoscopic Evaluation of Swallowing (FEES) is an instrumental assessment used to evaluate swallowing function. The Fiberoptic Endoscopic Dysphagia Severity Scale (FEDSS) is a tool used to rate the severity of dysphagia based on findings from FEES.
  The FEDSS ranges from Level 1 to Level 8, with Level 1 indicating normal swallowing physiology and Level 8 representing severe dysphagia with no protective laryngeal elevation. In this scale, a higher score indicates worse swallowing function, as higher levels indicate more severe dysphagia symptoms.
  The FEDSS is used to evaluate various aspects of swallowing function, including the efficiency of swallowing, the coordination between breathing and swallowing, and the presence of pharyngeal residue after swallowing. By identifying the severity of dysphagia using the FEDSS, clinicians can develop appropriate treatment plans to improve swallowing function and reduce the risk of complications.
Murray secretion scale | day 1, day 15, day 29, day 169
  The Murray secretion scale is a commonly used tool to assess the amount and characteristics of respiratory secretions in patients with respiratory diseases or conditions.
  It consists of a scoring system ranging from 0 to 4, with 0 indicating no secretions and 4 indicating thick, copious, and tenacious secretions that cannot be cleared.
  The scale assesses the color, amount, and viscosity of respiratory secretions, as well as the ease with which they can be cleared. The scale can be useful in monitoring the effectiveness of treatments aimed at reducing sputum production and improving airway clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Study Chair — Site Coordinator of United Medical Group
Locations (1):
- Xinzhu Rehabilitation Hospital, Xinzhu, Taiwan

IPD SHARING:
Plan to Share IPD: No